CLINICAL TRIAL: NCT06398808
Title: A Randomised, Double Blind, Parallel, Interventional Phase IIa Proof of Concept Trial to Evaluate the Efficacy and Safety of ZYIL1 for the Treatment of Patients With Mild to Moderately Active Ulcerative Colitis Resistant or Intolerant to Oral Aminosalicylates
Brief Title: A Study to Evaluate the Efficacy and Safety of ZYIL1 Oral Capsules for the Treatment of Patients With Mild to Moderately Active Ulcerative Colitis Resistant or Intolerant to Oral Aminosalicylates
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZYIL1.23.001
Record Dates: First submitted 2024-02-08; First posted 2024-05-03 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — 26S proteasome non-ATPase regulatory subunit 13; DMAC2L protein, human

STUDY DESIGN:
Intervention Model Description: randomly assigned in a 1:1 ratio
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (ZYIL1 capsules & placebo) (Active Comparator): ZYIL1 capsules 25 mg for oral administration + 50 mg placebo
  Interventions: Drug: Arm1
- Arm 2 (ZYIL1 capsules & placebo) (Active Comparator): ZYIL1 capsules 50 mg for oral administration + 25 mg placebo
  Interventions: Drug: Arm 2

INTERVENTIONS:
Drug: Arm1 — ZYIL1 capsules 25 mg for oral administration + 50 mg placebo
  Arms: Arm 1 (ZYIL1 capsules & placebo)
Drug: Arm 2 — ZYIL1 capsules 50 mg for oral administration + 25 mg placebo
  Arms: Arm 2 (ZYIL1 capsules & placebo)

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of ZYIL1 oral capsule twice a day for 12 weeks for treatment of mild to moderate active ulcerative colitis resistant or intolerant to oral aminosalicylates.

DETAILED DESCRIPTION:
This is a Phase IIa, randomized, two arms, double blind, double dummy, parallel, multicentre study to evaluate efficacy and safety of ZYIL1 oral capsules for the treatment of mild to moderately active ulcerative colitis resistant or intolerant to oral aminosalicylates.

The study consists

The study consists of: screening period of upto 4 weeks, treatment period of 12 weeks (first 6 weeks period: Induction period and remaining 6 weeks: Maintenance period), and end of the study at Week 13. The total duration of the study will be 119 days including screening period of 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 to 75 years, both inclusive.
2. Have had ulcerative colitis (UC) diagnosed at least 3 months prior to screening. The diagnosis of UC must be confirmed by endoscopic and histologic evidence.
3. Mild to Moderate active disease defined as total score of at least 4 on the mMS, endoscopy subscore of at least 2 and a rectal bleeding sub-score of at least 1.
4. Demonstrated an inadequate response to, loss of response to, or intolerance to any of the Oral aminosalicylates (e.g., mesalamine, sulfasalazine, olsalazine, balsalazide)

   ○ Signs and symptoms of persistently active disease, in the opinion of the investigator, during a current or prior course of at least 4 weeks of treatment with 2.4 g/day mesalamine, 4 g/day sulfasalazine, 1 g/day olsalazine, or 6.75 g/day balsalazide.
5. Have undergone colonoscopy within the past 2 years for extent of disease, and if the UC has been present for > 10 years, have had a colonoscopy with biopsy to rule out dysplasia
6. Patients who meet following laboratory values (assessed within 28 days prior to randomization):

   1. WBCs ≥2000/μL
   2. Neutrophils ≥1500/μL
   3. Platelets ≥100 X 10³/μL
   4. Hemoglobin ≥8.5 g/dL
   5. Serum creatinine of ≤1.5 X ULN or creatinine clearance >40 mL/minute (using Cockcroft/Gault formula)
   6. AST & ALT ≤1.5 X ULN
   7. Total bilirubin ≤ 1.5 X ULN
7. Men and women of childbearing potential must agree to use adequate birth control measures during the study. Acceptable methods of birth control in this study include: surgical sterilization, intrauterine device, oral contraceptive, contraceptive patch, long acting injectable contraceptive, partner's vasectomy, double-barrier method (condom or diaphragm with spermicide) or abstinence for at least 4 weeks prior to study drug administration, during study participation and for 30 days after their last dose of study drug.
8. All patients aged 45 years or over must have had a colonoscopy to screen for adenomatous polyps within 5 years of screening or must have had a colonoscopy at screening to assess for polyps.
9. Ability to provide written informed consent and to be compliant with the schedule of protocol assessments. In case of illiterate patients, thumb impression of the patients will be obtained along with the signature of the impartial witness or legally authorized representative (LAR) on the consent form prior to patient's participation in the trial.

Exclusion Criteria:

1. Diagnosis of Crohn's disease or indeterminate colitis or the presence or history of a fistula consistent with Crohn's disease.
2. Have severe extensive colitis as evidenced by at least one of the following:

   1. Physician judgment that the patient is likely to require colectomy or ileostomy within 12 weeks of baseline.
   2. Current evidence of fulminant colitis, toxic megacolon or bowel perforation.
   3. Previous total colectomy
   4. Have 4 or more of the following i.e Body temperature > 38 C,HR > 110 (bpm),Focal severe or rebound abdominal tenderness,Anemia (hemoglobin [Hgb] < 8.5 g/dL), Transverse colon diameter > 5 cm on plain X-ray.
3. Have positive stool culture for pathogens (O P, bacteria) or positive test for C.

   difficile at screening. If C. difficile is positive, the patient may be treated and retested.
4. Patients who have an evidence of pathogenic bowel infection.
5. History of recurrent or chronic infection (e.g. hepatitis B or C, syphilis, TB).
6. Laboratory test positive for HBsAg, HCV or HIV at screening.
7. Have had treatment with cyclosporine, tacrolimus, sirolimus, or mycophenolate mofetil (MMF) within 16 weeks of screening.
8. History or planned concurrent treatment with biological agents (infliximab, adalimumab, vedolizumab, and ustekinumab), immunosuppressive agents (e.g., azathioprine, 6-MP, or methotrexate) or with lymphocyte-depleting therapies (e.g., Campath, anti-CD4, cladribine, rituximab, ocrelizumab, cyclophosphamide, mitoxantrone, total body irradiation, bone marrow transplantation, alemtuzumab, daclizumab), Janus kinase (JAK) inhibitor (e.g.,Tofacitininb), steroids (e.g., prednisolone) prior to randomization.
9. History of treatment with an investigational agent within 5 half-lives of that agent prior to randomization.
10. History of treatment with topical rectal 5-ASA or steroids within 2 weeks of screening.
11. Receipt of a live vaccine within 4 weeks prior to randomization.
12. Chronic use of therapies that strongly inhibit or induce CYP3A4 metabolism within 4 weeks prior to randomization.
13. Clinically relevant cardiovascular, hepatic, neurological, pulmonary, ophthalmological, endocrine, psychiatric or other major systemic disease making implementation of the protocol or interpretation of the study difficult or that would put the patient at risk by participating in the study.
14. Pregnant or lactating women or women of child bearing potential who have positive serum beta HCG test at screening.
15. History of significant alcoholism or drug abuse within the past 1 year. History or presence of significant smoking (more than 10 cigarettes per day) or consumption of tobacco/nicotine products (more than 10 times per day).
16. History of difficulty with donating blood
17. Participants who have participated in any drug research study other than the present trial within past 3 months
18. Patients that have undergone significant trauma or major surgery within 4 weeks of screening visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of ZYIL1 for induction of clinical remission | Baseline to week 6
  clinical remission defined as an mMS score of 0 to 2, including: stool frequency subscore 0 or 1, rectal bleeding subscore 0 and endoscopy score 0 or 1.
  mMS;modified Mayo Score Minimum value "0" and Maxium Value "9" Higher scores means worse outcome compare to baseline.

SECONDARY OUTCOMES:
Proportion of participants achieving clinical response | Week 6 and Week 12
  Clinical Response defined decrease from baseline* in the mMS of greater than or equal to 2 points
  mMS;modified Mayo Score Minimum value "0" and Maxium Value "9" Higher scores means worse outcome compare to baseline.
Proportion of participants in clinical remission | Week 12
  clinical remission defined as an mMS score of 0 to 2, including: stool frequency subscore 0 or 1, rectal bleeding subscore 0 and endoscopy score 0 or 1.
  mMS;modified Mayo Score Minimum value "0" and Maxium Value "9" Higher scores means worse outcome compare to baseline.
Proportion of participants in endoscopic remission | Week 6 and Week 12
Mean change in biomarker fecal calprotectin | Baseline to Week 6 & Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Deven Parmar, MD,FCP, Study Chair — Zydus Therapeutics Inc.
Locations (1):
- ICON Hospital, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No